CLINICAL TRIAL: NCT00329537
Title: Open-Label Phase 1 Study to Assess the Tolerability, Pharmacokinetics and Safety of 2 and 6 µg/kg Sargramostim (SH L 04023) Administered Subcutaneously Once Daily for 4 Weeks, and Randomized, Double-Blind, Placebo-Controlled Phase 2 Study to Assess the Efficacy and Safety of 6 µg/kg Sargramostim (SH L 04023) Administered Subcutaneously Once Daily for 8 Weeks in Patients With Active Crohn's Disease (Sargramostim Phase 1/2 Study)
Brief Title: Study of Sargramostim in Moderately to Severely Active Crohn's Disease
Status: Terminated | Phase: Phase 2 | Type: Interventional
Sponsor: Genzyme, a Sanofi Company (Industry)
Responsible Party: Sponsor
Organization: Sanofi (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 309240; 91510
Record Dates: First submitted 2006-05-23; First posted 2006-05-24 (Estimated); Last update posted 2013-12-04 (Estimated); Status verified 2013-12

CONDITIONS: Crohn's Disease
Keywords: Crohn's Disease; Sargramostim; CDAI; Moderately to severely active Crohn's Disease
MeSH Terms: conditions — Crohn Disease | interventions — sargramostim

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Arm 1 (Experimental)
  Interventions: Drug: Sargramostim (Leukine)
- Arm 2 (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Sargramostim (Leukine) — Self-subcutaneous injection
  Other Names: BAY86-5326
  Arms: Arm 1
Drug: Placebo — Self-subcutaneous injection
  Arms: Arm 2

SUMMARY:
The purpose of this study is to assess the tolerability, pharmacokinetics and safety of 2 and 6 micro g/kg/day sargramostim administered subcutaneously once daily for 4 weeks, and to assess the efficacy and safety of 6 micro g/kg/day sargramostim administered subcutaneously once daily for 8 weeks in comparison with placebo, in patients with moderately to severely active Crohn's disease.

DETAILED DESCRIPTION:
On 29 May 2009, Bayer began transitioning the sponsorship of this trial to Genzyme. NOTE: This study was originally posted by sponsor Berlex, Inc. Berlex, Inc. was renamed to Bayer HealthCare, Inc.

ELIGIBILITY:
Inclusion Criteria:

* Confirmed diagnosis of Crohn's disease (endoscopic or radiological evaluation) at least 4 months prior to receiving the first dose of study drug
* Moderately to severely active Crohn's disease at time of screening (i.e., Crohn's disease activity index [CDAI] >220 and <475 points)

Exclusion Criteria:

* Colostomy or ileostomy
* Immediate need for gastrointestinal (GI) surgery for active GI bleeding, peritonitis, intestinal obstruction, or intra-abdominal or perianal abscess requiring surgical drainage
* GI surgery within 6 months prior to receiving the 1st dose of study drug
* Symptoms of bowel obstruction or confirmed evidence of a clinically-significant stricture within the last 6 months that has not been surgically corrected

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 11 (Actual)
Dates: Start 2006-06; Primary Completion 2007-05 (Actual); Study Completion 2007-05 (Actual)

PRIMARY OUTCOMES:
CDAI [Crohn's Disease Active Index] improvements | Baseline, 1w, 2w, 4w, 6w, 8w, 10w, 12w

SECONDARY OUTCOMES:
PRO [Patient-reported outcome] variables (QOL [Quality of life] | Baseline, 1w, 4w, 8w, 12w
PGI-C [Patient global impression of change]) | Baseline, 1w, 2w, 4w, 6w, 8w, 10w, 12w

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Genzyme, a Sanofi Company